CLINICAL TRIAL: NCT03402217
Title: Patient Centered Postpartum Contraception App
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: IRB17-12541
Record Dates: First submitted 2018-01-05; First posted 2018-01-18 (Actual); Results first posted 2024-05-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Contraceptive Usage
Keywords: Contraception; Post Partum Contraception
MeSH Terms: conditions — Contraception Behavior

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Patient Centered Postpartum Contraception App — This is a theory-based smart phone-based application designed to provide immediate postpartum contraception information to young women aged 15-25.

SUMMARY:
This study will evaluate a smart phone-based application ("app") designed to inform pregnant women ages 15-25 about their contraception options. The goal of this research will be to evaluate the usability, feasibility and acceptability of this app.

DETAILED DESCRIPTION:
This study will evaluate a smart phone-based application ("app") designed to inform pregnant women ages 15-25 about their contraception options. The goal of this research will be to evaluate the usability, feasibility and acceptability of this app. Participants will be asked to complete a survey after informed consent and before using the app. After using the app, participants will complete a second survey. This second survey will ask questions about the app including the following topics: Usability, user-friendliness, navigation, user interface, time spent, organization readability; Feasibility, informative, helpful, comprehensible, quality of art, interface, sound; and Acceptability breadth of content, depth of content, engaging and motivating, Innovative utility and value. Women will also rate the degree to which they promote use of the product: would use the app if available, believe the app will support contraceptive use and would recommend the app to peers. Study participation will end once participants are done with the second survey.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant
* Identify as African American or Black
* English as primary language

Exclusion Criteria:

* Not pregnant
* Not identifying as African American or Black
* Language other than English as primary language

Ages: 15 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: -Recruitment will occur at local primary care clinics.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-05-18 (Actual); Primary Completion 2019-01-07 (Actual); Study Completion 2019-01-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Gilliam, MD, MPH, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All recruitment was performed in clinic waiting rooms from May 2018-January 2019.
Pre-assignment Details: All enrolled participants were assigned to the single intervention group.
Groups:
- Single Arm Intervention Group: This is a single-arm pre-post study. The intervention group received the app intervention.
Period: Overall Study
Arm/Group | Single Arm Intervention Group
Started | 20
Completed | 19
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm Intervention Group
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3
  Between 18 and 65 years | 17
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 21.5 [17 to 25]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 20
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Application
Description: Feasibility, acceptability and usability of application. Mean of each item is reported. Each item has a possible score of 1-5, 1 = strongly disagree; 5= strongly agree. Higher scores indicate a better results for all items except "I found the app too complex to understand," "I think I would need tech support to use this app," "I thought there was too much inconsistency in app," "I found the app cumbersome to use," and "I needed to learn a lot before I could get going," where a lower score is a better result.
Time Frame: Immediately post intervention
Population: One individual of the 20 total participants completed the pre-test and received the intervention but did not complete the post-test.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Single Arm Intervention Group
Number analyzed (Participants) | 19
units on a scale
  How much do you like the look of the app? | 4.47 (.70)
  How much do you like the app itself? | 4.52 (.70)
  How would you rate the overall quality of this app | 4.16 (.96)
  Likelihood of recommending app to friends | 4.26 (.81)
  Rating the overall quality of the visuals: number analyzed (Participants) | 18
  Rating the overall quality of the visuals | 3.94 (1.35)
  Rating the overall quality of the audio | 4.42 (1.02)
  Rating the overall quality of the videos | 4.32 (.95)
  Information discussed was easy to understand | 3.58 (.96)
  Information discussed valuable to my repro health | 3.42 (1.02)
  Information helped me learn questions to ask Dr. | 4.32 (.95)
  I will use info provided by the app in the future. | 3.47 (.61)
  I can trust the info in the app. | 3.26 (.81)
  I would like to use this app frequently. | 3.05 (.85)
  I found the app too complex to understand. | 1.05 (1.31)
  I thought the app was easy to use. | 3.42 (.84)
  I think I would need tech support to use this app. | 1.05 (.74)
  I found the various functions were well-integrated | 3.0 (1.05)
  I thought there was too much inconsistency in app. | 1.15 (.89)
  Most people would learn to use app quickly. | 3.58 (.51)
  I found the app cumbersome to use. | 2.05 (1.58)
  I felt very confident using the app. | 3.42 (.69)
  I needed to learn a lot before I could get going. | 1.16 (1.21)

2. Secondary Outcome: Prior Method Use
Description: Methods of birth control participants have ever used
Time Frame: Pre-Survey
Measure: Number; unit: participants
Arm/Group | Single Arm Intervention Group
Number analyzed (Participants) | 20
participants
  Never used a birth control method | 3
  Withdrawal | 6
  Condoms | 11
  Oral contraceptive pill | 6
  Contraceptive ring | 1
  Contraceptive patch | 3
  Contraceptive injection | 11
  IUD | 0
  Implant | 2

3. Secondary Outcome: Number of Pregnancies (Including Current)
Time Frame: Pre-Survey
Measure: Median (Full Range); unit: events
Arm/Group | Single Arm Intervention Group
Number analyzed (Participants) | 20
events | 2 [1 to 4]

4. Secondary Outcome: Contraception Knowledge
Description: 7 questions assessing participant knowledge of different contraception methods
Time Frame: Pre-Survey
Measure: Mean (Standard Deviation); unit: correct answers
Arm/Group | Single Arm Intervention Group
Number analyzed (Participants) | 20
correct answers | 3.35 (1.14)

5. Secondary Outcome: Patient Activation
Description: Participant total of 13 Likert-style questions asking about how active a role they have taken in determining their health care. Measurement presented is the sum of 13 Likert items 1-5 to create a scale score. Possible score range from 13-65, with higher scores indicating more activation.
Time Frame: Pre-Survey, immediately post intervention
Population: as for outcome 1
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Single Arm Intervention Group
Number analyzed (Participants) | 19
score on a scale
  Pre-intervention | 62.0 (5.68)
  Post-intervention | 62.5 (6.27)
Statistical Analysis 1: Comparison: Single Arm Intervention Group; Pre and post-score paired comparison; Test type: Superiority; p = .383, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Information, Motivation and Behavioral Skills
Description: 15 questions asking participants about the information, motivation, and behavioral skills they possess relating to spacing pregnancies by 18 months or longer, split into information, motivation, and behavioral self-efficacy variables. Three subscales are presented: information subscale, motivation subscale, and behavioral skills subscale. The information scale is the summed correct answers to 7 questions, possible score 0-7. Motivation subscale is the sum of 6 Likert-type items with values from 1-4, for possible scores of 6-24; higher score is better. Behavioral skills subscale is the sum of 5 Likert-type items with values from 1-5, for possible subscales scores of 5-25; higher score is better.
Time Frame: immediately post intervention
Population: as for outcome 1
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Single Arm Intervention Group
Number analyzed (Participants) | 19
score on a scale
  Information pretest | 4.0 (1.69)
  Information posttest | 6.0 (1.18)
  Motivation pretest | 20.0 (2.52)
  Motivation posttest | 21.0 (2.41)
  Behavior pretest | 22.0 (3.45)
  Behavior posttest | 23.0 (3.27)
Statistical Analysis 1: Comparison: Single Arm Intervention Group; Information pre-post paired comparison; Test type: Superiority; p = .001, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Single Arm Intervention Group; Motivation pre- and post-paired comparison; Test type: Superiority; p = .07, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Single Arm Intervention Group; Behavior pre and post paired comparison; Test type: Superiority; p = .230, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Number of Children
Time Frame: Pre-Survey
Measure: Median (Full Range); unit: Children
Arm/Group | Single Arm Intervention Group
Number analyzed (Participants) | 20
Children | 1 [0 to 3]

8. Secondary Outcome: Number of Induced Abortions
Description: Previous miscarriages, abortions, times pregnant and children participants have
Time Frame: Pre-Survey
Measure: Median (Full Range); unit: Abortions
Arm/Group | Single Arm Intervention Group
Number analyzed (Participants) | 20
Abortions | 0 [0 to 1]

9. Secondary Outcome: Number of Miscarriages
Description: Previous miscarriages, abortions, times pregnant and children participants have
Time Frame: Pre-Survey
Measure: Median (Full Range); unit: Miscarriages
Arm/Group | Single Arm Intervention Group
Number analyzed (Participants) | 20
Miscarriages | 0 [0 to 2]

10. Other Pre Specified Outcome: Sociodemographic Information
Description: Monthly income
Time Frame: Pre-Survey
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm Intervention Group
Number analyzed (Participants) | 20
Participants
  Less than $500 | 6
  $500-999 | 9
  $1000-2000 | 3
  More than $2000 | 1
  No response | 1

ADVERSE EVENTS:
Time Frame: Duration of participation in the study (average 30 minutes per participant).
Description: This is a health education intervention and as such no adverse medical events were anticipated.
Arm/Group | Single Arm Intervention Group
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

LIMITATIONS AND CAVEATS:
Difficulty with recruiting eligible participants from clinic waiting rooms led to lower enrollment numbers than initially planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-07): https://cdn.clinicaltrials.gov/large-docs/17/NCT03402217/Prot_SAP_000.pdf